CLINICAL TRIAL: NCT02129192
Title: Bioequivalence of Telmisartan 80 mg/Amlodipine 5 mg/Hydrochlorothiazide 12.5 mg Fixed-dose Combination Tablet Compared to Concomitant Administration of Telmisartan 80 mg/Hydrochlorothiazide 12.5 mg Fixed-dose Combination Tablet and Amlodipine 5 mg Capsule in Healthy Male Subjects (an Open-label, Randomised, Single-dose, Two-sequence, Four-period Replicated Crossover Study), With Influence of Food on the Bioavailability of Telmisartan 80 mg/Amlodipine 5 mg/Hydrochlorothiazide 12.5 mg Fixed-dose Combination Tablet
Brief Title: Bioequivalence Study of Telmisartan Between Telmisartan 80 mg/Amlodipine 5 mg/Hydrochlorothiazide 12.5 mg (T80/A5/H12.5 mg) Fixed-dose Combination (FDC) Tablet and T80/H12.5 mg Tab and A5 mg (Encap A2.5 mg Tab x2) Concomitant Use
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1348.4
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Healthy
MeSH Terms: interventions — Amlodipine

ARMS (2):
- T80/A5/H12.5 mg FDC (Experimental): Telmisartan 80 mg/Amlodipine 5 mg/Hydrochlorothiazide 12.5 mg fixed dose combination tablet
  Interventions: Drug: T80/A5/H12.5 mg FDC tablet
- T80/H12.5 FDC + A5 mono (Active Comparator): Telmisartan 80 mg/Hydrochlorothiazide 12.5 mg fixed dose combination tablet and Amlodipine 5 mg capsule
  Interventions: Drug: Amlodipine 5mg capsule; Drug: T80/H12.5 mg FDC tablet

INTERVENTIONS:
Drug: Amlodipine 5mg capsule — Amlodipine 5mg capsule
  Arms: T80/H12.5 FDC + A5 mono
Drug: T80/H12.5 mg FDC tablet — Telmisartan 80 mg/Hydrochlorothiazide 12.5 mg FDC tablet
  Arms: T80/H12.5 FDC + A5 mono
Drug: T80/A5/H12.5 mg FDC tablet — Telmisartan 80 mg/Amlodipine 5 mg/Hydrochlorothiazide 12.5 mg FDC tablet
  Arms: T80/A5/H12.5 mg FDC

SUMMARY:
To investigate the steady state pharmacokinetics of different formulation of Telmisartan, Amlodipine, and Hydrochlorothiazide (HCTZ).

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects age >=20 and <=35 years; body weight: >=50 kg and <=80 kg; body mass index: >=18.0 and <=25.0 kg/m2
* Without any clinically significant findings and complications on the basis of a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR), body temperature)
* Signed and dated written informed consent prior to admission to the trial in accordance with the Good Clinical Practice (GCP) and the local legislation

Exclusion criteria:

- Any finding of the medical examination (including BP, PR and ECGs) deviating from normal and of clinical relevance

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Boehringer Ingelheim Investigational Site, Tokyo, Hachioji, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence TRRTT: Subjects were treated with telmisartan 80 mg (T80), amlodipine 5 mg (A5) and hydrochlorothiazide (HCTZ) 12.5 mg (H12.5 mg) in the following order from period 1 to period 5:
  T (test product: T80/A5/H12.5 mg fixed dose combination (FDC) tablet) - R (reference products: T80/H12.5 mg FDC tablet and A5 mg capsule) - R - T - T.
  Treatment periods 1 to 4 were administered following an overnight fast of at least 10 hours, in treatment period 5 after an overnight fast of at least 10 hours, a Japanese-style breakfast was served 30 minutes before drug administration
- Sequence RTTR: Subjects were treated telmisartan 80 mg (T80), amlodipine 5 mg (A5) and hydrochlorothiazide (HCTZ) 12.5 mg (H12.5 mg) in the following order from period 1 to period 4:
  R - T - T - R.
  The treatments were administered following an overnight fast of at least 10 hours.
Period: Period 1 Including Washout Period
Arm/Group | Sequence TRRTT | Sequence RTTR
Started | 36 | 36
Completed | 36 | 35 (Withdrawal by one subject in washout period)
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2 Including Washout Period
Arm/Group | Sequence TRRTT | Sequence RTTR
Started | 36 | 35
Completed | 36 | 35
Not Completed | 0 | 0
Period: Period 3 Including Washout Period
Arm/Group | Sequence TRRTT | Sequence RTTR
Started | 36 | 35
Completed | 36 | 35
Not Completed | 0 | 0
Period: Period 4 Including Washout Period
Arm/Group | Sequence TRRTT | Sequence RTTR
Started | 36 | 35
Completed | 36 | 35
Not Completed | 0 | 0
Period: Period 5
Arm/Group | Sequence TRRTT | Sequence RTTR
Started | 36 | 0 (This sequence consists of only 4 periods.)
Completed | 36 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This subject set included all subjects who were dispensed the study drug and were documented to have taken at least one dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence TRRTT | Sequence RTTR | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.6 (4.2) | 26.6 (3.9) | 26.6 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Maximum Measured Concentration (Cmax) of the Analytes in Plasma
Description: Maximum measured concentration (Cmax) of telmisartan, amlodipine and HCTZ in plasma
Time Frame: 3 hours (h) pre drug admin and 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 32h, 48h after drug admin, in addition 15min, 30min, 45min, 1h 30min, 2h 30min for telmisartan and HCTZ only, 72h for telmisartan and amlodipine only and 96h, 120h, 144h for amlodipine only
Population: Pharmacokinetic set (PKS) which included all healthy subjects in the TS who had evaluable PK variables for both treatments (i.e. had data of at least one analyte for both test and reference products) in periods 1, 2, 3 and 4. Subjects who had an important protocol violation relevant to PK evaluation were to be excluded from the PKS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- T80/H12.5 FDC + A5 Capsule: Telmisartan 80 mg/Hydrochlorothiazide 12.5 mg fixed dose combination tablet and Amlodipine 5 mg capsule
Arm/Group | T80/A5/H12.5 mg FDC | T80/H12.5 FDC + A5 Capsule
Number analyzed (Participants) | 71 | 71
ng/mL
  Telmisartan | 697 (75.5) | 726 (74.9)
  Amlodipine | 3.62 (20.2) | 3.57 (19.9)
  HCTZ | 98.5 (25.1) | 96.6 (25.8)
Statistical Analysis 1: Comparison: T80/A5/H12.5 mg FDC vs T80/H12.5 FDC + A5 Capsule; Adjusted by-treatment means on the log-transformed scale for telmisartan 80 mg; Test type: Non-Inferiority or Equivalence — Bioequivalence was established by using the average bioequivalence method and by ensuring that the ratio of Cmax of the two treatments was within the pre-specified acceptance range (80%-125%); Mixed Models Analysis; Model on logarithmic scale included "subjects within sequence" as random effect and "sequence", "period", and "treatment" as fixed effects; Adjusted geometric mean ratio (%) = 95.77, 90% CI 2-sided [88.89 to 103.17] — Ratio calculated as T80/A5/H12.5 mg FDC divided by T80/H12.5 FDC + A5 mono
Statistical Analysis 2: Comparison: T80/A5/H12.5 mg FDC vs T80/H12.5 FDC + A5 Capsule; Adjusted by-treatment means on the log-transformed scale for amlodipine 5 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 101.40, 90% CI 2-sided [99.70 to 103.13] — Ratio calculated as T80/A5/H12.5 mg FDC divided by T80/H12.5 FDC + A5 mono
Statistical Analysis 3: Comparison: T80/A5/H12.5 mg FDC vs T80/H12.5 FDC + A5 Capsule; Adjusted by-treatment means on the log-transformed scale for hydrochlorothiazide 12.5 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 101.77, 90% CI 2-sided [98.46 to 105.19] — Ratio calculated as T80/A5/H12.5 mg FDC divided by T80/H12.5 FDC + A5 mono

2. Primary Outcome: Maximum Measured Concentration (Cmax) of the Analytes in Plasma After Single Administration of T80/A5/H12.5 mg FDC Tablet
Description: Maximum measured concentration (Cmax) of telmisartan, amlodipine and HCTZ in plasma after single oral administration of T80/A5/H12.5 mg FDC tablet
Time Frame: as for outcome 1
Population: Food effect analysis set (FEAS) which included healthy subjects of treatment sequence TRRTT in the TS who were judged appropriate to continue to period 5 by the investigator, had evaluable PK variables for both feeding conditions and did not have an important protocol violation relevant to relative bioavailability evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- T80/A5/H12.5 mg FDC Fed: Telmisartan 80 mg/Amlodipine 5 mg/Hydrochlorothiazide 12.5 mg fixed dose combination tablet in fed condition
- T80/A5/H12.5 FDC Fasted: Telmisartan 80 mg/Amlodipine 5 mg/Hydrochlorothiazide 12.5 mg fixed dose combination tablet in fasted condition
Arm/Group | T80/A5/H12.5 mg FDC Fed | T80/A5/H12.5 FDC Fasted
Number analyzed (Participants) | 36 | 36
ng/mL
  Telmisartan | 182 (75.9) | 605 (84.4)
  Amlodipine | 3.54 (20.6) | 3.60 (22.4)
  HCTZ | 75.4 (16.5) | 94.6 (20.1)
Statistical Analysis 1: Comparison: T80/A5/H12.5 mg FDC Fed vs T80/A5/H12.5 FDC Fasted; Adjusted by-treatment geometric means for telmisartan 80 mg. No hypothesis was tested; Test type: Superiority or Other; p = 1.0000, ANOVA; Model included "subject" as random effect and "feeding condition" as fixed effect; Adjusted geometric mean ratio (%) = 30.15, 90% CI 2-sided [24.99 to 36.38] — Ratio calculated as T80/A5/H12.5 mg FDC Fed divided by T80/A5/H12.5 mg FDC Fasted
Statistical Analysis 2: Comparison: T80/A5/H12.5 mg FDC Fed vs T80/A5/H12.5 FDC Fasted; Adjusted by-treatment geometric means for amlodipine 5 mg. No hypothesis was tested; Test type: Superiority or Other; p < 0.0001, ANOVA; Model included "subject" as random effect and "feeding condition" as fixed effect; Adjusted geometric mean ratio (%) = 98.23, 90% CI 2-sided [94.63 to 101.97] — Ratio calculated as T80/A5/H12.5 mg FDC Fed divided by T80/A5/H12.5 mg FDC Fasted
Statistical Analysis 3: Comparison: T80/A5/H12.5 mg FDC Fed vs T80/A5/H12.5 FDC Fasted; Adjusted by-treatment geometric means for hydrochlorothiazide 12.5 mg. No hypothesis was tested; Test type: Superiority or Other; p = 0.5422, ANOVA; Model included "subject" as random effect and "feeding condition" as fixed effect; Adjusted geometric mean ratio (%) = 79.69, 90% CI 2-sided [74.97 to 84.71] — Ratio calculated as T80/A5/H12.5 mg FDC Fed divided by T80/A5/H12.5 mg FDC Fasted

3. Primary Outcome: Area Under the Concentration-time Curve (AUC 0-tz) of the Analytes in Plasma Over the Time Interval From 0 to the Last Quantifiable Plasma Concentration
Description: Area under the concentration-time curve (AUC 0-tz) of telmisartan, amlodipine and HCTZ in plasma over the time interval from 0 to the last quantifiable plasma concentration
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | T80/A5/H12.5 mg FDC | T80/H12.5 FDC + A5 Capsule
Number analyzed (Participants) | 71 | 71
ng*h/mL
  Telmisartan | 2580 (76.8) | 2600 (76.1)
  Amlodipine | 159 (23.4) | 157 (24.0)
  HCTZ | 600 (21.0) | 598 (19.1)
Statistical Analysis 1: Comparison: T80/A5/H12.5 mg FDC vs T80/H12.5 FDC + A5 Capsule; Adjusted by-treatment means on the log-transformed scale for telmisartan 80 mg; Test type: Non-Inferiority or Equivalence — Bioequivalence was established by using the average bioequivalence method and by ensuring that the ratio of AUC 0-tz of the two treatments was within the pre-specified acceptance range (80%-125%); Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 99.21, 90% CI 2-sided [96.14 to 102.38] — Ratio calculated as T80/A5/H12.5 mg FDC divided by T80/H12.5 FDC + A5 mono
Statistical Analysis 2: Comparison: T80/A5/H12.5 mg FDC vs T80/H12.5 FDC + A5 Capsule; Adjusted by-treatment means on the log-transformed scale for amlodipine 5 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 101.43, 90% CI [99.84 to 103.04] — Ratio calculated as T80/A5/H12.5 mg FDC divided by T80/H12.5 FDC + A5 mono
Statistical Analysis 3: Comparison: T80/A5/H12.5 mg FDC vs T80/H12.5 FDC + A5 Capsule; Adjusted by-treatment means on the log-transformed scale for hydrochlorothiazide 12.5 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 100.33, 90% CI 2-sided [98.29 to 102.40] — Ratio calculated as T80/A5/H12.5 mg FDC divided by T80/H12.5 FDC + A5 mono

4. Primary Outcome: Area Under the Concentration-time Curve (AUC 0-tz) of the Analytes in Plasma Over the Time Interval From 0 to the Last Quantifiable Plasma Concentration After Single Administration of T80/A5/H12.5 mg FDC Tablet
Description: Area under the concentration-time curve (AUC 0-tz) of telmisartan, amlodipine and HCTZ in plasma over the time interval from 0 to the last quantifiable plasma concentration after single administration of T80/A5/H12.5 mg FDC tablet
Time Frame: as for outcome 1
Population: FEAS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | T80/A5/H12.5 mg FDC Fed | T80/A5/H12.5 FDC Fasted
Number analyzed (Participants) | 36 | 36
ng*h/mL
  Telmisartan | 1500 (98.3) | 2350 (93.6)
  Amlodipine | 156 (23.9) | 157 (26.1)
  HCTZ | 515 (18.9) | 575 (19.2)
Statistical Analysis 1: Comparison: T80/A5/H12.5 mg FDC Fed vs T80/A5/H12.5 FDC Fasted; Adjusted by-treatment geometric means for telmisartan 80 mg. No hypothesis was tested; Test type: Superiority or Other; p = 1.0000, ANOVA; Model included "subject" as random effect and "feeding condition" as fixed effect; Adjusted geometric mean ratio (%) = 63.66, 90% CI 2-sided [58.98 to 68.71] — Ratio calculated as T80/A5/H12.5 mg FDC Fed divided by T80/A5/H12.5 mg FDC Fasted
Statistical Analysis 2: Comparison: T80/A5/H12.5 mg FDC Fed vs T80/A5/H12.5 FDC Fasted; Adjusted by-treatment geometric means for amlodipine 5 mg. No hypothesis was tested; Test type: Superiority or Other; p < 0.0001, ANOVA; Model included "subject" as random effect and "feeding condition" as fixed effect; Adjusted geometric mean ratio (%) = 99.74, 90% CI 2-sided [97.08 to 102.48] — Ratio calculated as T80/A5/H12.5 mg FDC Fed divided by T80/A5/H12.5 mg FDC Fasted
Statistical Analysis 3: Comparison: T80/A5/H12.5 mg FDC Fed vs T80/A5/H12.5 FDC Fasted; Adjusted by-treatment geometric means for hydrochlorothiazide 12.5 mg. No hypothesis was tested; Test type: Superiority or Other; p = 0.0001, ANOVA; Model included "subject" as random effect and "feeding condition" as fixed effect; Adjusted geometric mean ratio (%) = 89.66, 90% CI 2-sided [85.80 to 93.70] — Ratio calculated as T80/A5/H12.5 mg FDC Fed divided by T80/A5/H12.5 mg FDC Fasted

5. Secondary Outcome: Area Under the Concentration-time Curve (AUC 0-infinity) of the Analytes in Plasma Over the Time Interval From 0 to Extrapolated Infinity
Description: Area under the concentration-time curve (AUC 0-infinity) of telmisartan, amlodipine and HCTZ in plasma over the time interval from 0 to extrapolated infinity
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | T80/A5/H12.5 mg FDC | T80/H12.5 FDC + A5 Capsule
Number analyzed (Participants) | 71 | 71
ng*h/mL
  Telmisartan ( N = 142, 142) | 2750 (79.2) | 2730 (73.7)
  Amlodipine ( N = 142, 142) | 172 (25.4) | 170 (26.0)
  HCTZ ( N = 141, 142) | 626 (20.2) | 624 (18.2)
Statistical Analysis 1: Comparison: T80/A5/H12.5 mg FDC vs T80/H12.5 FDC + A5 Capsule; Adjusted by-treatment means on the log-transformed scale for telmisartan 80 mg; Test type: Non-Inferiority or Equivalence — Bioequivalence was established by using the average bioequivalence method and by ensuring that the ratio of AUC 0-inf of the two treatments was within the pre-specified acceptance range (80%-125%); Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 99.62, 90% CI 2-sided [96.32 to 103.04] — Ratio calculated as T80/A5/H12.5 mg FDC divided by T80/H12.5 FDC + A5 mono
Statistical Analysis 2: Comparison: T80/A5/H12.5 mg FDC vs T80/H12.5 FDC + A5 Capsule; Adjusted by-treatment means on the log-transformed scale for amlodipine 5 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 101.21, 90% CI 2-sided [99.59 to 102.87] — Ratio calculated as T80/A5/H12.5 mg FDC divided by T80/H12.5 FDC + A5 mono
Statistical Analysis 3: Comparison: T80/A5/H12.5 mg FDC vs T80/H12.5 FDC + A5 Capsule; Adjusted by-treatment means on the log-transformed scale for hydrochlorothiazide 12.5 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 100.15, 90% CI 2-sided [98.23 to 102.10] — Ratio calculated as T80/A5/H12.5 mg FDC divided by T80/H12.5 FDC + A5 mono

6. Secondary Outcome: Area Under the Concentration-time Curve (AUC 0-infinity) of the Analytes in Plasma Over the Time Interval From 0 to Extrapolated Infinity After Single Administration of T80/A5/H12.5 mg FDC Tablet
Description: Area under the concentration-time curve (AUC 0-infinity) of telmisartan, amlodipine and HCTZ in plasma over the time interval from 0 to extrapolated infinity after single administration of T80/A5/H12.5 mg FDC tablet
Time Frame: as for outcome 1
Population: FEAS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | T80/A5/H12.5 mg FDC Fed | T80/A5/H12.5 FDC Fasted
Number analyzed (Participants) | 36 | 36
ng*h/mL
  Telmisartan ( N = 35, 36 ) | 1670 (108.0) | 2530 (98.3)
  Amlodipine ( N = 36, 36 ) | 168 (26.0) | 169 (28.6)
  HCTZ ( N = 36, 36 ) | 542 (18.3) | 603 (18.3)
Statistical Analysis 1: Comparison: T80/A5/H12.5 mg FDC Fed vs T80/A5/H12.5 FDC Fasted; Adjusted by-treatment geometric means for telmisartan 80 mg. No hypothesis was tested; Test type: Superiority or Other; p = 1.0000, ANOVA; Model included "subject" as random effect and "feeding condition" as fixed effect; Adjusted geometric mean ratio (%) = 64.40, 90% CI 2-sided [59.59 to 69.59] — Ratio calculated as T80/A5/H12.5 mg FDC Fed divided by T80/A5/H12.5 mg FDC Fasted
Statistical Analysis 2: Comparison: T80/A5/H12.5 mg FDC Fed vs T80/A5/H12.5 FDC Fasted; Adjusted by-treatment geometric means for amlodipine 5 mg. No hypothesis was tested; Test type: Superiority or Other; p < 0.0001, ANOVA; Model included "subject" as random effect and "feeding condition" as fixed effect; Adjusted geometric mean ratio (%) = 99.45, 90% CI 2-sided [96.69 to 102.29] — Ratio calculated as T80/A5/H12.5 mg FDC Fed divided by T80/A5/H12.5 mg FDC Fasted
Statistical Analysis 3: Comparison: T80/A5/H12.5 mg FDC Fed vs T80/A5/H12.5 FDC Fasted; Adjusted by-treatment geometric means for hydrochlorothiazide 12.5 mg. No hypothesis was tested; Test type: Superiority or Other; p < 0.0001, ANOVA; Model included "subject" as random effect and "feeding condition" as fixed effect; Adjusted geometric mean ratio (%) = 89.82, 90% CI 2-sided [86.02 to 93.79] — Ratio calculated as T80/A5/H12.5 mg FDC Fed divided by T80/A5/H12.5 mg FDC Fasted

ADVERSE EVENTS:
Time Frame: From first drug administration until end of washout period (14 days) or 144 hours after last drug administration (6 days)
Groups:
- Total.: All participants randomised into the study.
Arm/Group | T80/A5/H12.5 mg FDC | T80/H12.5 FDC + A5 Capsule | Total.
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 11/71 | 6/72 | 16/72
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T80/A5/H12.5 mg FDC (N=71) | T80/H12.5 FDC + A5 Capsule (N=72) | Total. (N=72)
Headache (Nervous system disorders) | 7 | 4 | 10
Orthostatic hypotension (Vascular disorders) | 4 | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.